CLINICAL TRIAL: NCT02567422
Title: A Phase I Study of M6620 (VX-970, Berzosertib) in Combination With Cisplatin and XRT in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC; SDC 10060121)
Brief Title: Testing the Addition of M6620 (VX-970, Berzosertib) to Usual Chemotherapy and Radiation for Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01643; NCI-2015-01643 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9950 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 9950 (Other: CTEP); N01CM00100 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2025-06-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Carcinoma of Unknown Primary; Head and Neck Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage III Laryngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage III Sinonasal Squamous Cell Carcinoma AJCC v6 and v7; Stage IV Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IV Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IV Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Sinonasal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — berzosertib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (berzosertib, cisplatin, radiation therapy) (Experimental): Patients receive berzosertib IV over 60 minutes on day -7 and then weekly on day 2 and cisplatin IV over 30-60 minutes weekly on day 1. Patients also undergo radiation therapy once daily, 5 days a week. Treatment continues for up to 7 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT, PET/CT, or MRI throughout the study.
  Interventions: Drug: Berzosertib; Drug: Cisplatin; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of berzosertib (M6620) when given together with cisplatin and radiation therapy in treating patients with head and neck squamous cell carcinoma that has spread from where it started to nearby tissue or lymph nodes (locally advanced). M6620 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving M6620 together with cisplatin and radiation therapy may work better in treating patients with locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of M6620 (VX-970, berzosertib) when administered along with weekly cisplatin and radiation therapy (XRT) in patients with locoregionally advanced head and neck squamous cell carcinoma (HNSCC).

II. Establish the recommended phase 2 dose (RP2D) of the combination.

SECONDARY OBJECTIVES:

I. Characterize the pharmacokinetic (PK) profile of M6620 (VX-970, berzosertib).

II. Assess for potential drug-drug interaction between M6620 (VX-970, berzosertib) and aprepitant.

III. To observe and record anti-tumor activity. IV. To assess the rate of complete metabolic response (CMR) at 12 weeks post completion of chemoradiation using 18 fluorodeoxyglucose (FDG) positron emission tomography (PET) scans.

V. To collect archival tumor material for retrospective analysis of association between tissue-based biomarkers and clinical outcome.

OUTLINE: This is a dose-escalation study of berzosertib.

Patients receive berzosertib intravenously (IV) over 60 minutes on day -7 and then weekly on day 2 and cisplatin IV over 30-60 minutes weekly on day 1. Patients also undergo radiation therapy once daily, 5 days a week. Treatment continues for up to 7 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT), PET/CT, or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up for 30 days, every 2 weeks for 3 months, and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed head and neck squamous cell cancer (HNSCC) including paranasal sinus cancers but excluding nasopharyngeal carcinomas
* Clinical staged III or IV HNSCC, according to American Joint Committee on Cancer (AJCC) 7th Edition, that is not amenable to surgical resection
* Carcinoma of the neck of unknown primary site origin (regardless of HPV/p16 status) is eligible
* Age >= 18 years; because no dosing or adverse event data are currently available on the use of M6620 (VX-970, berzosertib) in combination with cisplatin in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of M6620 (VX-970, berzosertib) on the developing human fetus are unknown; for this reason and because DNA-damage response (DDR) inhibitors as well as other therapeutic agents used in this trial may have teratogenic potential, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months after completion of M6620 (VX-970, berzosertib) administration
* Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential who are sexually active should be willing and able to use medically acceptable forms of contraception throughout the treatment phase of the trial and for up to 6 months following the last administration of study treatment; men who are sexually active must be willing and able to use medically acceptable forms of contraception throughout the treatment phase of the trial and for 6 months after completion of M6620 (VX-970, berzosertib) administration

Exclusion Criteria:

* Patients with nasopharyngeal carcinoma, skin squamous cell carcinoma (SCC), and salivary gland carcinomas are not eligible
* Patients who are receiving adjuvant chemoradiation after surgical resection of the primary site of disease
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients on tacrolimus or any other immunosuppressants with significant interaction with cisplatin
* Patient who requires live vaccine administration
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX-970, berzosertib) or cisplatin
* Prior systemic chemotherapy for the current cancer (prior chemotherapy for a different cancer is allowed)
* Prior receipt of radiotherapy that would result in overlap of the new and old radiation therapy fields
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring intravenous antibiotics at the time of treatment initiation
  * Symptomatic congestive heart failure (requiring hospital stay within the last 6 months)
  * Myocardial infarction within the last 6 months
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because M6620 (VX-970, berzosertib) as a DNA-damage response (DDR) inhibitor may have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620 (VX-970, berzosertib), breastfeeding should be discontinued if the mother is treated with M6620 (VX-970, berzosertib); these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients with well-controlled disease, as determined by CD4 count and viral load, who are on antiretroviral therapy that does not contain a strong inducer or inhibitor of CYP3A4 are allowed on trial; HIV-positive patients on combination antiretroviral therapy with strong inducers or inhibitors of CYP3A4 are ineligible because of the potential for pharmacokinetic interactions; patients with poorly controlled HIV are not eligible due to the increased risk of lethal infections when treated with marrow-suppressive therapy
* Definitive clinical or radiographic evidence of distant metastasis or adenopathy below the clavicles
* M6620 (VX-970, berzosertib) is primarily metabolized by CYP3A4; therefore, concomitant administration with strong inhibitors or inducers of CYP3A4 should be avoided; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-05-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek K Owonikoko, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (19):
- United States (19):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Patients received M6620 (VX-970, berzosertib) 120 mg/m2 by infusion in their arm weekly, cisplatin 40 mg/m2 IV weekly starting a week after M6620, and radiation therapy 70 Gy daily Monday-Friday also starting a week after M6620.
- Dose Level 2: Patients received M6620 (VX-970, berzosertib) 160 mg/m2 by infusion in their arm weekly, cisplatin 40 mg/m2 IV weekly starting a week after M6620, and radiation therapy 70 Gy daily Monday-Friday also starting a week after M6620.
- Dose Level 3; Dose Level 3 Expansion: Patients received M6620 (VX-970, berzosertib) 200 mg/m2 by infusion in their arm weekly, cisplatin 40 mg/m2 IV weekly starting a week after M6620, and radiation therapy 70 Gy daily Monday-Friday also starting a week after M6620.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 3 Expansion
Started | 11 | 6 | 11 | 15
Completed | 11 | 6 | 11 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 3 Expansion | Total
Number analyzed (Participants) | 11 | 6 | 11 | 15 | 43
Age, Continuous [Median (Full Range); unit: Years] | 69 [49 to 76] | 65.5 [52 to 72] | 59 [50 to 75] | 59 [45 to 74] | 61 [45 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 5 | 17
  Male | 6 | 4 | 6 | 10 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 6 | 10 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 2 | 5
  White | 8 | 6 | 10 | 11 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 11 | 15 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Grade 3, 4, and 5 Adverse Events
Description: According to the Cancer Therapy Evaluation Program National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v. 5). The highest grade experienced by the participant will be reported.
Time Frame: Up to 6.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 3 Expansion
Number analyzed (Participants) | 11 | 6 | 11 | 15
Participants
  Grade 5 | 0 | 0 | 1 | 1
  Grade 4 | 3 | 3 | 4 | 3
  Grade 3 | 7 | 3 | 5 | 11
  Grades 1-2 | 1 | 0 | 1 | 0

2. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicities
Description: Dose limiting toxicities are protocol-specific adverse events considered at least possibly related to the study intervention. Graded according to NCI CTCAE v5.
Time Frame: Up to 3 weeks after completion of radiation therapy
Population: Dose limiting toxicities (DLTs) are only evaluated in participants during dose escalation (i.e. Dose Levels 1, 2, and 3). Participants not completing the treatment for reasons other than an adverse event (i.e. withdrawal or non-compliance with treatment) are excluded from the analysis. DLTs were not evaluated for participants enrolled in Dose Expansion.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 9 | 6 | 9
Participants
  Experiencing a DLT | 2 | 1 | 2
  Did not experience a DLT | 7 | 5 | 7

3. Primary Outcome: Establish the Recommended Phase 2 Dose (RP2D)
Description: Defined as the highest doses of cisplatin and berzosertib safely combined with radiation.
Time Frame: Up to 7 weeks
Measure: Number; unit: mg/m^2
Groups:
- Dose Escalation: Patients received different doses of M6620 (VX-970, berzosertib) by infusion in their arm weekly, cisplatin 40 mg/m2 IV weekly starting a week after M6620, and radiation therapy 70 Gy daily Monday-Friday also starting a week after M6620.
Arm/Group | Dose Escalation
Number analyzed (Participants) | 28
mg/m^2 | 200

4. Secondary Outcome: Pharmacokinetic Characteristics of Berzosertib
Description: The maximum concentration ratio between Day -7 collections to Day 2 collections. Collection time points are baseline, 30 and 55 minutes after the start of M6620 infusion, 5, 15, 30 minutes, 1, 2, 4, 23 (Day 3), 48 (Day 4), and 72 hours (Day 5) after the end of M6620 infusion given on Day 2.
Time Frame: Up to Day 5
Population: Based on samples collected. PK was only collected in the dose escalation phase. PK was not collected for participants in the dose expansion arm.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 5 | 0 | 5
ratio | 0.75 (1.7) |  | 1.02 (1.5)

5. Secondary Outcome: Potential Drug-drug Interaction
Description: The maximum concentration of M6620 in the blood when aprepitant is also given.
Time Frame: Up to Day 5
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 5 | 0 | 5
ug/L | 732 (2.5) |  | 1149 (1.9)

6. Secondary Outcome: Number of Participants Experiencing a Response
Description: Evaluated by Response Evaluation Criteria in Solid Tumors 1.1. Response is defined as complete response (disappearance of all target and non-target lesions) or partial response (at least a 30% decrease in the sum of diameters of target lesions from baseline).
Time Frame: Up to 6.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 3 Expansion
Number analyzed (Participants) | 11 | 6 | 11 | 15
Participants
  Response | 9 | 2 | 7 | 7
  No Response | 0 | 1 | 1 | 3
  Not Performed | 2 | 3 | 3 | 5

7. Secondary Outcome: Number of Participants Experiencing a Metabolic Response
Description: Assessed by fluorodeoxyglucose-positron emission tomography (FDG PET) and measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Metabolic response are participants demonstrating a complete response (disappearance of all target and non-target lesions) or a partial response (at least a 30% decrease in the sum of diameters of target lesions from baseline).
Time Frame: At week 12 after completing intervention
Population: Due to funding issues, response was solely assessed by CT scans instead of FDG PET. Metabolic data was therefore not collected.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Expression of Tissue-based Biomarkers as Markers of Deoxyribonucleic Acid Damage and Predictors of Clinical Outcome
Description: Kaplan-Meier curves for Progression Free Survival (PFS), defined as time to disease progression, and Overall Survival (OS), defined as time until death or off study, were used to evaluate if the gene expression profiles of ERCC1 and XRCC1, and TP53 correlated to these outcomes.
Time Frame: Up to 6.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 3 Expansion
Number analyzed (Participants) | 8 | 5 | 9 | 9
Participants
  Selected Biomarkers correlated to Outcome | 0 | 0 | 0 | 0
  Selected Biomarkers did not correlate to Outcome | 8 | 5 | 9 | 9

ADVERSE EVENTS:
Time Frame: Up to 6.5 years
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 3 Expansion
All-Cause Mortality (participants affected / at risk) | 2/11 | 1/6 | 2/11 | 2/15
Serious Adverse Events (participants affected / at risk) | 5/11 | 4/6 | 7/11 | 5/15
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6 | 11/11 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=11) | Dose Level 2 (N=6) | Dose Level 3 (N=11) | Dose Level 3 Expansion (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 0
Fever (General disorders) | 1 | 1 | 2 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
infections and infestations: positive blood culture (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 2 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pseudogout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=11) | Dose Level 2 (N=6) | Dose Level 3 (N=11) | Dose Level 3 Expansion (N=15)
Anemia (Blood and lymphatic system disorders) | 9 | 6 | 7 | 11
DVT (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 1
Heart racing (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 5
Ear fullness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 1 | 1 | 1
Heightened sense of hearing (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 4 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Vision changes' (Eye disorders) | 0 | 0 | 1 | 0
Visual disturbance (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 1 | 7 | 7
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 6 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 3 | 7 | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 3 | 2
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth cavity erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth sores (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 1 | 7 | 12
Nausea (Gastrointestinal disorders) | 7 | 5 | 6 | 11
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 2 | 4 | 1 | 2
Thickened saliva (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Tongue swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 5
Chills (General disorders) | 2 | 1 | 1 | 0
Edema limbs (General disorders) | 2 | 1 | 4 | 3
Fatigue (General disorders) | 7 | 4 | 6 | 11
Fever (General disorders) | 1 | 2 | 1 | 1
Hemoptysis (General disorders) | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 1
Leg cramp (General disorders) | 0 | 1 | 0 | 0
Localized edema (General disorders) | 1 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 1
Neck edema (General disorders) | 0 | 1 | 1 | 0
Pain (General disorders) | 3 | 2 | 2 | 5
Post-op Delerium (General disorders) | 0 | 0 | 1 | 0
Soreness gum (General disorders) | 0 | 1 | 0 | 0
Soreness left side (General disorders) | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Aspiration pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 1
Candida Albicans (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1
Thrush (Infections and infestations) | 1 | 2 | 0 | 4
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 7 | 6 | 5 | 11
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Secretion from trach site (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Acute transminitis (Investigations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 4
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increase (Investigations) | 0 | 0 | 0 | 6
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 0
Creatinine decreased (Investigations) | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 4 | 0 | 2 | 0
GGT increased (Investigations) | 1 | 1 | 1 | 2
Lymphocyte count decreased (Investigations) | 7 | 4 | 7 | 11
Neutrophil count decreased (Investigations) | 5 | 3 | 5 | 7
Platelet count decreased (Investigations) | 7 | 4 | 7 | 10
Weight loss (Investigations) | 7 | 3 | 9 | 9
White blood cell decreased (Investigations) | 7 | 4 | 5 | 12
Anorexia (Metabolism and nutrition disorders) | 5 | 2 | 3 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1 | 3
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0 | 5 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 1 | 3 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 5 | 4 | 9
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3 | 4 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Cramping in R foot/ankle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 0 | 2 | 5
Dysgeusia (Nervous system disorders) | 6 | 4 | 6 | 8
Headache (Nervous system disorders) | 3 | 1 | 3 | 2
Hyperosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Lightheadedness (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 1 | 0
Subjective diminished fine motor control (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Xtrapyramidal disorder: restless legs (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 3
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 5
Sputum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Allodynia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Erythema of buccal mucosa (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Excoriations around PEG tube insertion site (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Radiation mucositis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1
Redness and local irritation at G tube site (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Skin manifestations (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Sores on chin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
PEG tube placement (Surgical and medical procedures) | 2 | 0 | 0 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 3 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Lymphedema (Vascular disorders) | 0 | 1 | 0 | 2
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02567422/Prot_SAP_000.pdf